CLINICAL TRIAL: NCT05719922
Title: Low-load Blood Flow Restriction Exercise Versus Conventional Heavier Load Resistance Training Exercise in UK Military Personnel With Persistent Knee Pain: A Multi-centre Randomized Controlled Trial
Brief Title: The ADAPTation to Therapeutic Resistance Training (ADAPT) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Defence Medical Rehabilitation Centre, UK (Other Government)
Collaborators: University of Bath (Other)
Responsible Party: Principal Investigator, Peter Ladlow, Higher Scientific Officer, Defence Medical Rehabilitation Centre, UK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DefenceMedRC
Record Dates: First submitted 2023-01-19; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Musculoskeletal Injury; Muscle Weakness
Keywords: Musculoskeletal rehabilitation; Blood flow restriction; Resistance training; knee pain; military
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-load blood flow restriction training (LL-BFR) (Experimental): Twice daily LL-BFR for 3 weeks
  Interventions: Other: Resistance Training
- Heavier load resistance training (HL-RT) (Active Comparator): Three sessions per week for 3 weeks
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Resistance Training — Comparing two different exercise-based treatment methodologies on the clinical outcomes of individuals with persistent knee pain.

SUMMARY:
In 2018, the Academic Department of Military Rehabilitation (ADMR) published a pilot randomised controlled trial (RCT), demonstrating the feasibility and acceptability of integrating twice-daily blood flow restriction (BFR) training into a busy residential care setting. Following its publication was a guidance note written by the Directorate of Defence Rehabilitation restricting the implementation of BFR training until more evidence can be provided to support its efficacy. This research trial is a fully-powered, multi-centre RCT investigating the efficacy and biological mechanism underpinning BFR therapy in UK military personnel with lower-limb musculoskeletal injury (specifically, persistent anterior knee pain) during residential rehabilitation. This study will aim to optimise both the rehabilitation outcome and improve the time-and cost-effectiveness of the service delivered across UK Defence Rehabilitation and beyond. Results will provide insight and knowledge to the clinical and scientific community to not only those embedded within Defence Rehabilitation, but also those working in civilian sector organisations and professional sport in the UK and abroad.

ELIGIBILITY:
Inclusion Criteria:

* mechanical knee pain for at least three months
* present with clinical signs and symptoms of knee pain arising from the tibiofemoral or patellofemoral joint diagnosed by sport and exercise medicine physician and/or physiotherapist
* have reduced occupational employability medical grade secondary to their knee pain
* report progression of resistance training load within the patient's rehabilitation programme is limited by knee pain
* aged between 18 and 55 years
* available to attend for the entire duration of the RRU course and a review appointment 3-months following course.

Exclusion Criteria:

diagnosed tibial, femoral or patella fracture and/or dislocation;

* present with instability in the knee resulting from ligament deficiency
* present with clinical signs and symptoms of patellar tendinopathy
* have planned surgery over the study period
* restricted knee range of movement; clinical signs and symptoms of non-musculoskeletal or serious pathological condition (i.e. Inflammatory arthropathy, infection or tumour) or referred pain from non-local pain source
* present with any physical impairment or co-morbidities (including cardio-vascular disease) precluding the safe participation in the rehabilitation programme and/or assessment procedures
* Cortico-steroid or analgesic injection intervention within the previous 7-days or previous knee surgery within the last 12 months to the affected limb

Medical Exclusion Criteria:

* History of cardiovascular disease including hypertension, peripheral vascular disease, thrombosis/embolism, ischaemic heart disease, myocardial infarction.
* History of the following musculoskeletal disorders: rheumatoid arthritis, avascular necrosis or osteonecrosis, severe osteoarthritis.
* History of the following neurological disorders: Peripheral neuropathy, Alzheimer's disease, amyotrophic lateral sclerosis, Parkinson's disease, severe traumatic brain injury.
* Varicose veins in the lower limb
* Acute viral or bacterial upper or lower respiratory infection at screening
* Known or suspected lower limb chronic exertional compartment syndrome (CECS)
* Postsurgical swelling
* Surgical insertion of metal components at the position of cuff inflation
* History of any of the following conditions or disorders not previously listed: diabetes, active cancer
* History of elevated risk of unexplained fainting or dizzy spells during physical activity/exercise that causes loss of balance
* History of haemorrhagic stroke or exercise induced rhabdomyolysis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Extremity Functional Scale (LEFS) over time | Baseline, week 3 and week 15
  LEFS is a 20-question patient-reported outcome measure (PROM) that measures functional status in patients with lower limb musculoskeletal injury. Questions on activity vary in physical demand from walking to running on uneven ground. The LEFS is a validated tool and has demonstrated good test-retest reliability and responsiveness in individuals with persistent knee pain.

SECONDARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) over time | Baseline, week 3 and week 15
Change in Patient Specific Functional Scale over time | Baseline, week 3 and week 15
Change in Musculoskeletal Health Questionnaire (MSK-HQ) over time | Baseline, week 3 and week 15
Change in Tampa Scale of Kinesiophobia (TSK) over time | Baseline, week 3 and week 15
Health Anxiety Depression Scale (HADS) | Baseline
Change in International Physical Activity Questionnaire (IPAQ) over time | Baseline, week 3 and week 15
Change in Numeric Pain Rating Scale (NPRS) over time | Baseline, week 3 and week 15
Change in Sport Injury Rehabilitation Beliefs Survey (SIRBS) over time | Baseline, week 3 and week 15
Change in functional Activity Assessment (FAA) over time | Baseline and week 15
Change in five Repetition Maximum Leg Press over time | Baseline, week 3 and week 15
Change in isometric muscle strength of hip and knee using hand-held dynamometer over time | Baseline, week 3 and week 15
Change in single leg heel raises to fatigue over time | Baseline, week 3 and week 15
Change in qualitative assessment of single leg squat (QASLS) over time | Baseline, week 3 and week 15
Change in decline knee bend over time | Baseline, week 3 and week 15
Change in isometric midthigh pull over time | Baseline, week 3 and week 15
Change in counter-movement jump over time | Baseline, week 3 and week 15
Change in knee extension and flexion - maximal isometric voluntary contraction over time | Baseline, week 3 and week 15
Change in muscle volume and anatomical cross sectional area (CSA) using magnetic resonance imaging (MRI) over time | Baseline, week 3 and week 15
Change in pennation angle over time using ultrasonography | Baseline, week 3 and week 15
  Pennation angle measured in degrees
Change in fascicle length over time using ultrasonography | Baseline, week 3 and week 15
  fascicle length measured in mm
Change in single leg squat over time - kinetic and kinematic analysis | Baseline, week 3 and week 15
  3D motion capture and force plate data will be used to collect kinetic and kinematic data which will be later analysed using inverse dynamics. Force measured in Newtons, Moments measured in Newton/Metres/kg
Change in bilateral squat over time - kinetic and kinematic analysis | Baseline, week 3 and week 15
  3D motion capture and force plate data will be used to collect kinetic and kinematic data which will be later analysed using inverse dynamics. Force measured in Newtons, Moments measured in Newton/Metres/kg
Change in markers of muscle damage over time | Baseline, week 3 and week 15
  Using fasted blood samples. E.g., Creatine Kinase (units/L)
Change in markers of oxidative stress over time | Baseline, week 3 and week 15
  Using fasted blood samples. E.g., Protein carbonyl (units/L)
Change in markers of inflammation over time | Baseline, week 3 and week 15
  Using fasted blood samples. E.g., Interleukin-6 (pg/ml)
Change in markers of endothelial function over time | Baseline, week 3 and week 15
  Using fasted blood samples. E.g., Vascular endothelial growth factor (µg/L)
Change in daily monitoring of wellness score over time | Daily for the 3 weeks of rehabilitation
  Subjective patient reported outcome measure of 'wellness' scored using a 5-point likert scale.
Change in daily monitoring of session rate of perceived exertion (sRPE) over time | Daily for the 3 weeks of rehabilitation
  Subjective patient reported outcome measure of exertion, scored 0 to 10 (0 = no exertion, 10= maximal exertion)
Change in daily monitoring of pain over time | Daily for the 3 weeks of rehabilitation
  Subjective patient reported outcome measure of pain measured using a 0 to 100mm visual analog scale (VAS). 0= no pain, 100 = worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bennett, PhD, Study Chair — Defence Medical Rehabilitation Centre
Locations (6):
- United Kingdom (6):
  - RRU Aldershot, Aldershot
  - RRU Colchester, Colchester
  - RRU Cranwell, Cranwell
  - RRU Edinburgh, Edinburgh
  - RRU St Athan, St Athan
  - RRU Bulford, Tidworth

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be made available upon reasonable request to the chief investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the dissemination of research findings (i.e, publications and conference proceedings)
Access Criteria: Most data will be openly available but, due to privacy concerns, some data regarding participants are available only to bona fide researchers working on a related project, subject to the completion of a non-disclosure agreement.

REFERENCES:
- [Derived] Cassidy RP, Lunt KM, Coppack RJ, Bennett AN, Bilzon JLJ, Mcguigan MP, Egginton N, Sellon E, Day J, Ladlow P. ADAPTations to low load blood flow restriction exercise versus conventional heavier load resistance exercise in UK military personnel with persistent knee pain: protocol for the ADAPT study, a multi-centre randomized controlled trial. BMC Musculoskelet Disord. 2023 Jul 17;24(1):580. doi: 10.1186/s12891-023-06693-3. PMID 37461024